CLINICAL TRIAL: NCT06087536
Title: A Prospective, Multinational, Multicenter, Randomized, Sequential, Double-blind, Placebo-controlled, Phase 2a Clinical Trial to Assess the Safety and Pharmacokinetics of OMN6 in HABP or VABP Caused by Acinetobacter Baumannii Complex (ABC).
Brief Title: A Clinical Trial to Assess the Safety and PK of OMN6 in HABP or VABP Caused by Acinetobacter Baumannii Complex
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Omnix Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: OMN6-002
Record Dates: First submitted 2023-07-25; First posted 2023-10-17 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Hospital-acquired Bacterial Pneumonia; Ventilator-associated Bacterial Pneumonia
Keywords: HABP VABP ABC Acinetobacter baumannii pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OMN6 treatment (Experimental): OMN6 on top of Meropenem and Colistin
  Interventions: Drug: OMN6
- Placebo (Placebo Comparator): Placebo on top of Meropenem and Colistin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OMN6 — Cohort 1: 50 mg x 3/day Cohort 2: 100 mg x 3/day Cohort 3: 150 mg x 3/day
  3 x 3-hour IV infusions for 1 Day of treatment concomitant with background antimicrobial treatment with meropenem plus colistin for 7 to 14 days
  Arms: OMN6 treatment
Drug: Placebo — 3 x 3-hour IV infusions for 1 Day of treatment concomitant with background antimicrobial treatment with meropenem plus colistin for 7 to 14 days
  Arms: Placebo

SUMMARY:
This is a phase 2a, multinational, multicenter, double-blind, randomized, placebo-controlled, dose-ranging safety, tolerability and PK study in patients with HABP (Hospital Acquired Bacterial Pneumonia) or VABP (Ventilator Associated Bacterial Pneumonia) caused by ABC to identify safe and well-tolerated doses and to assess the PK profile of OMN6 in patients.

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent form.
2. Male or female patients 18 years or older
3. A diagnosis of either a HABP or a VABP
4. ABC infection of the lower respiratory tract suspected based on a positive rapid testing of respiratory specimens
5. Women of childbearing potential (WOCBP) (i.e., not post-menopausal or surgically sterilized) must have a negative highly sensitive urine or serum pregnancy test before randomization.
6. Acute Physiology and Chronic Health Evaluation II (APACHE II) score between 10 and 24

Exclusion Criteria:

1. Moderate to severe reduction of renal function
2. Liver dysfunction
3. Evidence of septic shock
4. Acute respiratory distress syndrome.
5. Immunosuppressed patients (due to either immunosuppressant drugs or to any medical condition).
6. History of any known hypersensitivity to colistin or to carbapenems
7. Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of the study data

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of a single-day treatment with OMN6 vs. matching placebo when coadministered with a background therapy of meropenem and colistin | 28 day
  Incidence of TEAE and SAEs by frequency, severity, relatedness, and outcome, clinical laboratory findings change from baseline, vital signs and ECGs change from baseline.
To asses the Cmax of OMN6 in patient population | 1 day
  Maximum Observed Plasma Concentration
To assess the Tmax of OMN6 in patient population | 1 day
  Time to Cmax
To assess the AUC of OMN6 in patient population | 1 day
  Area Under the Plasma Concentration-Time Curve
To assess the t1/2 of OMN6 in patient population | 1 day
  Time to Half-life

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Omnix Medical Research Site, Be’er Ya‘aqov
  - Omnix Medical Research Site, Holon
  - Omnix Medical Research Site, Petah Tikva
  - Omnix Medical Research Site, Rishon LeZiyyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: OMN6 a novel bioengineered peptide for the treatment of multidrug resistant Gram negative bacteria — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7988117/
- See also: In Vitro and In Vivo Antimicrobial Activity of the Novel Peptide OMN6 against Multidrug-Resistant Acinetobacter baumannii — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9494975/